CLINICAL TRIAL: NCT02410538
Title: Frequently Asked Questions as an Help to Improve the Information of ICU Patients' Families.
Brief Title: Frequently Asked Questions for ICU Patients' Families
Acronym: FamiréaXVII
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_3678
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-04

CONDITIONS: Improve the Understanding of the Diagnosis the Treatment and the Prognosis by One Member of the Family

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- families that received the list of "FAQ": The intervention consists of the delivery to the relatives of ICU patients a list of "21 key issues" in intensive care during the first 48h period of ICU stay, only for intubated and mechanically ventilated patients A formal interview is scheduled to relatives of ICU patients on D3 of inclusion
  Interventions: Other: list of "FAQ"
- families that received information as usual: A formal interview is scheduled relatives of ICU patients on D3 inclusion
  Interventions: Other: list of "FAQ"

INTERVENTIONS:
Other: list of "FAQ"

SUMMARY:
The intervention consists of the delivery of a list of 21 questions to the relative of each patient admitted in ICU, intubated and mechanically ventilated during the first 48 hours of the stay. A formal interview is scheduled for relatives at Day 3 of inclusion. The information comprehension at Day 5 (± 1) will be compared between families that received the list of "FAQ" and families that received information as usual (without providing the list of FAQ

DETAILED DESCRIPTION:
Half of the families of ICU patients do not understand the information provided by doctors and nurses. Receiving clear, loyal and appropriate information is one of their main expectations. We have previously reported that relatives had difficulty asking questions that allow them to improve their understanding regarding ICU issues. In a preliminary study, we developed a list of questions considered as important by families, ICU doctors and nurses.

The aim of this prospective, randomized and controlled trial is to test the effectiveness of a list of frequently asked questions to relatives of ICU patients on their understanding of the provided information.

The intervention consists of the delivery of a list of 21 questions to the relative of each patient admitted in intensive care, intubated and mechanically ventilated in the first 48 hours of ICU stay. A formal interview is scheduled for relatives at Day 3 of inclusion. The information comprehension at Day 5 (± 1) will be compared between families that received the list of "FAQ" and families that received information as usual (without providing the list of FAQ).

ELIGIBILITY:
Inclusion Criteria:

The subjects that will be included are relatives of patients. The patients must be

1. Adults
2. Receiving invasive mechanical ventilation
3. Intubated in the first 48 hours of ICU admission
4. For an expected duration of mechanical ventilation > 48 hours
5. With a life expectancy of at least 5 days and a SAPS 2 at baseline < 75
6. Who received a visit within 24 hours after intubation. Only one relative will be included.

Exclusion Criteria:

* person unable to read French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: relative of each patient admitted in intensive care, intubated and mechanically ventilated in the first 48 hours of the stay.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of understanding at day 5 by a method of reformulation questionnaire | 5th day after inclusion
  The physician in charge of the patient provides the diagnosis, the treatment and the prognosis to the investigator prior to meet the relative. After the meeting, the relative gives to the investigator the diagnosis, main treatements and the prognosis as they have undestood them.
  In a final step, the investigator will indicate whether similar responses are consistent or not consistent.
Scale of satisfaction out of intensive care. | 3 months and at one yearfter inclusion
  HADS scores and IES-R at day 5 to day 10.

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hôpital Nord Assistance Publique Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Azoulay E, Forel JM, Vinatier I, Truillet R, Renault A, Valade S, Jaber S, Durand-Gasselin J, Schwebel C, Georges H, Merceron S, Cariou A, Moussa M, Hraiech S, Argaud L, Leone M, Curtis JR, Kentish-Barnes N, Jouve E, Papazian L. Questions to improve family-staff communication in the ICU: a randomized controlled trial. Intensive Care Med. 2018 Nov;44(11):1879-1887. doi: 10.1007/s00134-018-5423-2. Epub 2018 Oct 21. PMID 30374690